CLINICAL TRIAL: NCT01634919
Title: A Single Center, Prospective Study Evaluating the Anti-fibrotic Effect of Combination Therapy of Peginterferon Alpha-2a Plus Ribavirin in Patients with Chronic Hepatitis C, Based on Histologic Changes and Noninvasive Fibrosis Assessments
Brief Title: Histologic Changes and Noninvasive Assessment in Hepatitis C Patients Treated with Peginterferon Alpha-2a and Ribavirin
Status: Completed | Type: Observational
Sponsor: Seoul National University Boramae Hospital (Other)
Responsible Party: Principal Investigator, Won Kim, MD, PhD, Assistant Professor, Seoul National University Boramae Hospital
Other Study IDs: 06-2012-74
Record Dates: First submitted 2012-07-03; First posted 2012-07-06 (Estimated); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic hepatitis C; Liver fibrosis; ARFI(Acoustic radiation force impulse)
MeSH Terms: conditions — Hepatitis C, Chronic; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Liver tissue in frozen states
  * Whole blood including PBMC and sera
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic hepatitis C: Chronic hepatitis C
  Interventions: Device: chronic hepatitis C

INTERVENTIONS:
Device: chronic hepatitis C — acoustic radiation force impulse ultrasonography
  Other Names: noninvasive fibrosis imaging

SUMMARY:
•The purpose of this study is to compare the performance between liver biopsy and non-invasive fibrosis assessments evaluating anti-fibrotic efficacy of peginterferon plus ribavirin in patients with hepatitis C pre- and post-treatment

DETAILED DESCRIPTION:
* Patients with histologically advanced hepatitis C receiving peginterferon plus ribavirin combination therapy have showed 30-40% of a sustained virologic response (SVR) rate and 50% of histologic improvement.
* The histologic change of liver is the most important prognosticator to predict further clinical outcomes in advanced hepatitis C patients following peginterferon-based antiviral therapy.
* Although liver biopsy remains the gold standard for histologic assessment, it has several shortcomings in terms of poor repeatability due to its invasiveness and poor reproducibility due to sampling error and intra- or inter-observer variability.
* Treatment-naïve patients with chronic hepatitis C will receive PEGASYS® 180 mcg once weekly and ribavirin twice daily for 24 or 48 weeks depending on the genotype of hepatitis C virus (HCV).
* All subjects will be followed for up to 48 weeks after treatment cessation.
* Liver biopsy will be done at baseline and the end of follow-up for the evaluation of histologic response.
* Noninvasive tests for liver fibrosis (ARFI elastography, APRI, FIB-4, FibroTest®, and ELF test) will be assessed per 24 weeks during the whole study period.
* The results of this study will provide insight into the histo-physical link between histologic changes and liver stiffness dynamics during and after peginterferon alpha-2a plus ribavirin treatment in patients with advanced hepatitis C.
* Therefore, noninvasive fibrosis assessments may be useful to trace fibrosis outcomes in patients with advanced hepatitis C receiving antiviral therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects ≥20 years of age
* Subjects with positive anti-HCV Ab in sera
* Subjects with detectable HCV RNA by quantitative real time polymerase chain reaction (PCR) (> 50 IU/mL)
* Subjects without receiving any previous antiviral treatment
* Subjects undergoing radiologic studies (liver ultrasonography (USG), CT or MRI) to exclude the presence of hepatocellular carcinoma (HCC) within the last 1 year before enrolment
* All fertile males with partners of childbearing age and females must be using reliable contraception during the study and for 3 months after treatment completion
* Written informed consent should be obtained from all subjects.

Exclusion Criteria:

* History of any interferon (IFN)-based therapy before enrolment
* Positive test at screening for anti-hepatitis A virus (HAV) immunoglobulin M (IgM) Ab, HBsAg, anti-hepatitis D virus (HDV) Ab or anti- HIV Ab
* Histologically confirmed liver cirrhosis (F4 of fibrosis stage)
* If subjects have compromised liver function (Child-Pugh score >6)
* Signs or symptoms of hepatocellular carcinoma within the last 1 year before enrolment
* History or other evidence of a medical condition associated with chronic liver disease other than viral hepatitis (e.g., hemochromatosis, autoimmune hepatitis, metabolic liver disease, alcoholic liver disease, toxin exposures, thalassemia)
* Women with ongoing pregnancy or who are breast feeding
* Male partner of potentially pregnant women
* Neutrophil count <1,500 cells/mm3 or platelet count <75,000 cells/mm3 at screening
* Hemoglobin <11 g/dL for females and <12 g/dL for men at screening
* Serum creatinine level >1.5 times the upper limit of normal at screening
* Evidence of immunosuppressive therapy
* History of severe psychiatric disease, especially depression.(Severe psychiatric disease is defined as major depression or psychosis, suicidal attempt, hospitalization for psychiatric disease, or a period of disability due to a psychiatric disease)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital-based cohort
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2012-07; Primary Completion 2017-02-17 (Actual); Study Completion 2018-02-09 (Actual)

PRIMARY OUTCOMES:
Anti-fibrotic response | 48 weeks after the end of treatment
  Anti-fibrotic response, indicated by a lack of histological worsening, defined as the stabilization or the improvement of at least one stage in the histologic fibrosis staging 48 weeks after the end of treatment

SECONDARY OUTCOMES:
Histologic and noninvasive fibrosis assessments | 48 weeks after the end of treatment
  * Liver fibrosis score(according to the viral genotype or virologic response)
  * Morphometric analysis of fibrosis surface area
  * Acoustic radiation force impulse (ARFI) ultrasound imaging and clinical fibrosis indices (APRI, FIB-4, FibroTest®, and ELF test)
  * Noninvasive tests using the tissue shear wave speed and clinical fibrosis indices

CONTACTS AND LOCATIONS:
Overall Officials: Won Kim, Ph.D, Principal Investigator — SMG-SNU Boramae Medical Center
Locations (2):
- South Korea (2):
  - Seoul Metropolitan Government Boramae Medical Center, Seoul
  - SMG-SNU Boramae Medical Center, Seoul